CLINICAL TRIAL: NCT05088824
Title: When and Why Desarda Repair
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Boshra Nashaat, resident doctor, Assiut University
Other Study IDs: Desarda
Record Dates: First submitted 2021-09-24; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed with oblique inguinal hernia
  Interventions: Procedure: hernia repair by desarda technique

INTERVENTIONS:
Procedure: hernia repair by desarda technique — It involves use of undetached strip of external oblique aponeurosis to strengthen the posterior wall of the inguinal canal which is based on the physiological principles. This is a physiological repair and is tension free, can be used in strangulated hernia

SUMMARY:
One of the most significant subjects studied in abdominal wall surgery is inguinal hernia. Its management is very codified.

The main factors evaluating efficient hernia surgery are not only the rate of complications (recurrence and groin pain essentially) but also cost and time to return to normal activities.

Desarda technique is a non-mesh technique described first in 2001. This surgical technique uses a flap of external oblique aponeurosis in place of a mesh. Its singularity remains its low cost, no use of mesh, and less extensive dissection

Mesh repair has its own limitations; it is unphysiological as mesh is used. Chronic inguinal pain, seroma formation, foreign body sensation, risk of mesh infection are common complications and not recommended in strangulated hernias and extra cost involved by the mesh itself.

It involves use of undetached strip of external oblique aponeurosis to strengthen the posterior wall of the inguinal canal which is based on the physiological principles. This is a physiological repair and is tension free, can be used in strangulated hernia. Recurrence and complication rates equal to or less than Lichtenstein's repair. It's a simple procedure, early ambulation and less time of hospital stay, low cost for the patient as mesh is not used and most importantly no question of mesh related complications such as mesh rejection, infection, migration and foreign body sensation and chronic groin pain which is comparatively low in this procedure.

ELIGIBILITY:
Inclusion Criteria:

* primary inguinal hernia
* Aged 18 and above
* reducible inguinal or inguino-scrotal hernia

Exclusion Criteria:

* Obstructive uropathy or chronic obstructive pulmonary disease
* incarcerated hernia
* recurrent hernia
* bilateral hernia
* active infection at groin area
* pantalloon hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective clinical trial will be conducted on 30 patients diagnosed with oblique inguinal hernia . The study population will go for hernia repair by Desarda technique .
  The treatment will be herniorrhaphy. All the patients will be followed up after the 1st week, 1st month, 3 month and after 6 month . The efficacy and adverse effects will be compared by statistical analysis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
postoperative hospital stay | 6 month
  the duration of postoperative hospital stay
chronic pain | 6 months
  the patient will be assed for the presence of feeling of pain after the procedure or not
recurrence | 6 months
  the patient will be followed up for recurrence of hernia in the same place by clinical examination

IPD SHARING:
Plan to Share IPD: Undecided